CLINICAL TRIAL: NCT00734409
Title: Combining Objective and Subjective Sedation Assessment Tools - Second Study
Brief Title: Combining Objective and Subjective Sedation Assessment Tools
Acronym: COST_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00002117; DUHS parent 3930938 (Other Grant/Funding Number: Covidien)
Record Dates: First submitted 2008-06-03; First posted 2008-08-14 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-08

CONDITIONS: Critical Illness
Keywords: Mechanical ventilation; Human; conscious sedation; bispectral index; monitoring; critical care; propofol
MeSH Terms: conditions — Critical Illness | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RASS plus (BIS) (Experimental): Participants in this arm will receive sedation assessment with the RASS scale augmented with Bispectral Index (BIS) Monitor
  Interventions: Device: Bispectral Index (BIS) Monitor
- RASS only (No Intervention): Participants will receive sedation assessment only using the RASS scale which is the standard of care at our institution

INTERVENTIONS:
Device: Bispectral Index (BIS) Monitor — BIS monitoring in addition to RASS assessments
  Other Names: Richmond agitation sedation scale; neurofunction monitor
  Arms: RASS plus (BIS)

SUMMARY:
The purpose of this study is to determine if the use of a device called the BIS monitor in addition to the Richmond Agitation Sedation Scale will give better assessment of a subject's level of sedation.

DETAILED DESCRIPTION:
Patients in the intensive care unit (ICU) who require a ventilator to help them breathe also require sedation in order to keep them comfortable and prevent injury. The national guidelines for sedation management include a daily interruption of sedation performed once each morning. To determine the amount of sedation needed, the current standard practice is to use a system called the Richmond Agitation-Sedation Scale (RASS). The patient is stimulated by calling their name or by tapping their shoulder until the patient's responses indicate that a satisfactory level of sedation has been achieved.

The purpose of this study is to determine if the use of a device called the BIS monitor in addition to the RASS will give better assessment of a subject's level of sedation. The BIS monitor is a sensor strip taped to the forehead and attached to a device that reads electrical activity from the brain. It is approved by the U.S. Food and Drug Administration (FDA) for monitoring patients under sedation.

ELIGIBILITY:
Inclusion Criteria:

* patient in the ICU
* continuous IV sedation with propofol midazolam or dexmedetomidine
* age > 18
* expected to require mechanical ventilation for >=48 hours

Exclusion Criteria:

* prisoners
* no available space on forehead
* continuous electroencephalography(EEG) monitoring
* bifrontal brain injury
* barbiturate coma therapy
* known hypersensitivity to study medications
* high risk for ethanol (ETOH) withdrawal
* resuscitation from cardiac arrest without recovery of mental status
* moribund clinical state (death expected within 48 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-05; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, PhD RN, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were in the Medical ICU or Neuro ICU at Duke University Hospital or the mixed ICU at Durham Regional. If patients met all inclusion criteria and no exclusion criteria, the attending was asked if patient's legally authorized representative (LAR) could be approached for consent. Enrollment started May of 2008 and closed April of 2011.
Pre-assignment Details: Patients were only excluded from the trial after consent and prior to randomization if they no longer met inclusion criteria, for instance the medical team decided to remove sedatives.
Groups:
- RASS Plus BIS: Participants in this arm will receive sedation assessment with the RASS scale augmented with BIS monitoring.
Period: Overall Study
Arm/Group | RASS Plus BIS | RASS Only
Started | 155 | 145
Completed | 155 | 145
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RASS Plus BIS | RASS Only | Total
Number analyzed (Participants) | 155 | 145 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 102 | 99 | 201
  >=65 years | 53 | 46 | 99
Age Continuous [Mean (Standard Deviation); unit: years] | 53.95 (18.15) | 57.7 (15.30) | 55.78 (16.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 71 | 147
  Male | 79 | 74 | 153
Region of Enrollment [Number; unit: participants]
  United States | 155 | 145 | 300

OUTCOME MEASURES:

1. Primary Outcome: Mean Sedative Use
Description: The mean amount of propofol used on each patient while the patient was in the ICU and receiving mechanical ventilation.
Time Frame: Intensive Care Unit (ICU) stay through discharge
Population: All patients who met eligibility requirements, consented for the trial, and were randomized were included in the analysis.
Measure: Mean (Standard Deviation); unit: ml/hour
Arm/Group | RASS Plus BIS | RASS Only
Number analyzed (Participants) | 155 | 145
ml/hour | 13.35 (11.79) | 15.54 (11.88)

2. Secondary Outcome: Unplanned Self-device Removal Events
Description: The number of unplanned self-device removal events that took place during the study period.
Time Frame: ICU stay through discharge
Population: as for outcome 1
Measure: Number; unit: Event
Arm/Group | RASS Plus BIS | RASS Only
Number analyzed (Participants) | 155 | 145
Event | 0 | 1

3. Secondary Outcome: Mean Days on Mechanical Ventilation
Description: The mean number of days that the patients were on mechanical ventilation.
Time Frame: ICU stay- through discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RASS Plus BIS | RASS Only
Number analyzed (Participants) | 155 | 145
Days | 7.43 (8.32) | 6.85 (12.57)

ADVERSE EVENTS:
Arm/Group | RASS Plus BIS | RASS Only
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/145
Other Adverse Events (participants affected / at risk) | 0/155 | 1/145
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RASS Plus BIS (N=155) | RASS Only (N=145)
Unplanned Self-Device Removal Event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No